CLINICAL TRIAL: NCT00403741
Title: Effects of Individuals Consultations in Adapted Physical Activity on Behaviours in Physical Exercise by Type 2 Diabetics
Brief Title: Consultations in Adapted Physical Activity on Behaviours in Physical Exercise by Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: National Institut of Prevention and Health Education (Unknown)
Responsible Party: HALIMI Serge, Professor, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0621
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: behavior; physical activity; motivation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: motivational interviewing

SUMMARY:
Assesment the impact of three individuals consultations in adapted physical activity by type 2 diabetics

DETAILED DESCRIPTION:
Regular physical activity is now recognized for its beneficial effects on physiological and psychological characteristics of type 2 diabetic individuals.

However, initiating a physical activity program for type 2 diabetics strikes in practice to somatic and psychological obstacles which explain many results studies on compliance.

Instituting educational strategies in physical activity seems essential in order to provoke changes in patients' behaviours and to modify incompatible habits with the disease.

The main objective of for this study is to assess the impact of three individual consultations in Adapted Physical Activity (APA) on the self-determined motivation for physical exercise of type 2 diabetics. These three consultations will be proposed fifteen months after a therapeutic education session and based on the principles of motivational interviewing developed by Miller & Rollnick (2002).

The secondary objectives of this study are to assess the impact of these three consultations on other psychological (perceived competence in physical exercise, perceived support, quality of life, locus of control, health beliefs) and behavioural (Physical activity compliance, health condition) characteristics.

120 persons type 2 diabetics, aged between 18 and 80, will be recruited after the day which estimate the therapeutic education training proposed in the Department of Diabetic Education of Grenoble University Hospital. Two groups will randomized: 60 patients in experimental group and 60 patients in control group.

Self-determined motivation will be estimated by a french version of the Treatment Self-Regulation Questionnaire (TSRQ ; Ryan & Connell, 1989 ; Williams, Freedman & Deci, 1998).

Health behaviour compliance related to diabetic disease and its treatment will be assessed with the " revised Summary of Diabetes Self-Cares Activities " (SDSCA) (Toobert, Hampson, & Glasgow, 2000).

Perceived competence in physical exercise will be measured with a french version of the Perceveid Competence Diabetes Scale (PCDS) (Williams, Freedman & Deci, 1998).

Perceptions of autonomy, competence and relatedness support will be assessed with the Health Care Climate Quetionnaire (HCCQ) (Williams, Grow, Freedman, Ryan & Deci, 1996) and the Interpersonal Behaviours Scale (Otis & Pelletier, in press).

Patient's quality of life will be evaluated with the Diabetes Quality of Life (DQOL) adapted for type 2 diabetics by Senez, Felicciolo, Moreau and Le Goaziou (2004).

The locus control will be assessed with the Diabetes Locus of Control Scale (DLCS ; Pruyn et al., (1988; Watson et al., 1990).

The person's health condition will be measured by the HbA1c amount and the lipid profile (cholesterol, HDL, LDL, triglycerides)

Four times for estimations variables will be realized:

* Time 1 : the day which estimates the therapeutic education training
* Time 2 : + 3 mois
* Time 3 : + 9 mois
* Time 4 : + 15 mois The control group will receive therapeutic education training in Department Education Diabetic of the University Hospital of Grenoble and a "day test" (one day which estimate this training).

For the experimental group, three consultations in Adapted Physical Activity (APA) will be proposed after the "day test".

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetics
* age < 80 years
* to be able to read and to understand French
* to be affiliate national insurance
* to give a light and read consent

Exclusion Criteria:

* incapacity to carry out a questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Score on Treatment Self-Regulation Questionnaire(TSRQ)at Treatment Self-Regulation Questionnaire (TSRQ) at 3 months, 9 months and 15 months after assesment's day of the education period.

SECONDARY OUTCOMES:
Modifiable Activity Questionnaire(MAQ)at 3 months, 9 months and 15 months after assesment's day of the education period.
Perceveid Competence Scale (PCS)at assesment's day of the education period and at 3 months, 9 months and 15 months after assesment's day of the education period.
Interpersonal behaviors scale at assesment's day of the education period and at 3 months, 9 months and 15 months after assesment's day of the education period.
Diabetes Quality of Life (DQOL) at assesment's day of the education period and at 15 months after assesment's day of the education period.
Diabetes Locus of Control Scale (DLCS)at assesment's day of the education period and at 15 months after assesment's day of the education period.
HbA1c et lipid profile at 3 months, 9 months and 15 months after assesment's day of the education period.

CONTACTS AND LOCATIONS:
Overall Officials: HALIMI SH Serge, PU-PH, Principal Investigator — University Hospital, Grenoble